CLINICAL TRIAL: NCT06730685
Title: PHILUCA: The Development of Muscle Mass, Muscle Strength, and Muscle Function in Patients With Lung Cancer During Cancer Treatment
Brief Title: Sarcopenia and Cachexia in Patients With Lung Cancer
Acronym: PHILUCA
Status: Enrolling by invitation | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Susanne Dalton, Professor, MD, PhD, Zealand University Hospital
Other Study IDs: PHILUCA; SJ-1081 (Other: Research Ethics Committee Region Zealand)
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Small Cell Lung Cancer (SCLC)
Keywords: Sarcopenia; Cachexia; Treatment-tolerance; Survival; Quality of Life; Lung cancer; Muscle function; Muscle strength; Muscle mass
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Sarcopenia; Cachexia; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PHILICA study investigates whether muscle mass, muscle strength, and muscle function are associated with treatment tolerance, quality of life and survival in patients with lung cancer. It also aims to explore why some patients face challenges in completing their treatment. The findings may contribute to improved strategies for supporting patients and developing more precise and individualized treatment plans in the future.

DETAILED DESCRIPTION:
The PHILUCA prospective cohort study investigates the relationship between sarcopenia, cachexia, and change in muscle parameters with both treatment tolerance, quality of life and survival in patients with lung cancer receiving systemic treatment(s) (n=160). It aims to identify factors associated with difficulties in completing oncological treatment and to elucidate patterns that may inform improved patient support and individualized treatment planning. The study involves non-invasive physical assessments, patient-reported questionnaires, and the analysis of routinely collected medical data.

Assessments of muscle mass, muscle strength, muscle function, and quality of life are conducted at key time points, including at diagnosis and after three months into treatment or until the first control scan. Physical tests are performed during routine hospital visits, requiring no additional appointments. Body composition analysis is performed using Bioelectrical impedance analysis and by Computed Tomography scans obtained as part of standard care, without additional imaging procedures.

All participants receive standard lung cancer treatment, which may include surgery, chemotherapy, radiation therapy, immunotherapy, targeted therapy, or combinations thereof, based on disease type and stage. The study does not interfere with or modify standard care protocols. Participants unwilling or unable to fully participate may still contribute by completing a baseline questionnaire and consenting to the use of medical record data.

The study seeks to advance the understanding of how muscle-related parameters influence cancer treatment outcomes. The findings are anticipated to inform strategies for optimizing treatment tolerance, improving patient outcomes, and tailoring supportive care interventions for individuals with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Diagnosed with lung cancer (all types and stages) and scheduled for oncological treatment
* More than 3 months expected survival

Exclusion Criteria:

* Competing cancer
* Pregnancy
* Severe physical or cognitive disabilities preventing physical testing and informend consent
* Not able to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed and treated at Zealand University Hospital, Naestved Hospital
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Overvall survival | 12 months from inclusion
  Death from all causes

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLT) | 6 months from inclusion
  DLT defined as switching treatment; treatment delay (≥3 days from initially planned); treatment de-escalation (dose reduction ≥15% of platinum agent); early treatment termination; and hospitalization ≥1 day, all due to chemotherapy-induced side effects.
Haematological toxicities | 6 months from inclusion
  Anaemia; Leukocytopenia; Neutropenia; Thrombocytopenia. Graded by the Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0
Change in muscle mass | Assessments are intended to be performed around 3 months after inclusion, which in routine clinical practice usually corresponds to the time point immediately before the first control scan.
  Measured at the 3rd lumbar vertebrae. Routine CT-scans (from baseline CT to last performed CT)
Change in muscle function | Assessments are intended to be performed around 3 months after inclusion, which in routine clinical practice usually corresponds to the time point immediately before the first control scan.
  10 meter habitual and maximal gait speed (m/s)
Change in muscle function | Assessments are intended to be performed around 3 months after inclusion, which in routine clinical practice usually corresponds to the time point immediately before the first control scan.
  30-second sit to stand (5 x times sit to stand measured concurrently)
Change in muscle strength | Assessments are intended to be performed around 3 months after inclusion, which in routine clinical practice usually corresponds to the time point immediately before the first control scan.
  Maximal isometric handgrip strength by dynamometry
Health-Related Quality of Life | Assessments are intended to be performed around 3 months after inclusion, which in routine clinical practice usually corresponds to the time point immediately before the first control scan.
  Measured by the EORTC Questionnaire Core 30 (QLQ-C30). The QLQ-C30 questionnaire consists of 30 questions with five functional scales (physical, role, cognitive, emotional and social), three symptom scales, a global health status / QoL scale, and six single items.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Disease-specific symptoms | Assessments are intended to be performed around 3 months after inclusion, which in routine clinical practice usually corresponds to the time point immediately before the first control scan.
  Measured by the EORTC lung module (QLQ-LC13). The QLQ-LC13 module comprises both multi-item and single-item measures of lung cancer-associated symptoms (coughing, haemoptysis, dyspnoea and pain) and side-effects from conventional chemo- and radiotherapy (hair loss,neuropathy, sore mouth and dysphagia).
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Oksbjerg Dalton, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
For statistical analyses all data will be transferred to the Danish Cancer Institute
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning when data collection are finalized and ending 5 years after the publication of results

REFERENCES:
- [Background] Sayer AA, Cooper R, Arai H, Cawthon PM, Ntsama Essomba MJ, Fielding RA, Grounds MD, Witham MD, Cruz-Jentoft AJ. Sarcopenia. Nat Rev Dis Primers. 2024 Sep 19;10(1):68. doi: 10.1038/s41572-024-00550-w. PMID 39300120
- [Background] Dalton SO, Steding-Jessen M, Jakobsen E, Mellemgaard A, Osterlind K, Schuz J, Johansen C. Socioeconomic position and survival after lung cancer: Influence of stage, treatment and comorbidity among Danish patients with lung cancer diagnosed in 2004-2010. Acta Oncol. 2015 May;54(5):797-804. doi: 10.3109/0284186X.2014.1001037. Epub 2015 Mar 12. PMID 25761702
- [Background] Buentzel J, Heinz J, Bleckmann A, Bauer C, Rover C, Bohnenberger H, Saha S, Hinterthaner M, Baraki H, Kutschka I, Emmert A. Sarcopenia as Prognostic Factor in Lung Cancer Patients: A Systematic Review and Meta-analysis. Anticancer Res. 2019 Sep;39(9):4603-4612. doi: 10.21873/anticanres.13640. PMID 31519557
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Srdic D, Plestina S, Sverko-Peternac A, Nikolac N, Simundic AM, Samarzija M. Cancer cachexia, sarcopenia and biochemical markers in patients with advanced non-small cell lung cancer-chemotherapy toxicity and prognostic value. Support Care Cancer. 2016 Nov;24(11):4495-502. doi: 10.1007/s00520-016-3287-y. Epub 2016 May 28. PMID 27236439
- [Background] Sjoblom B, Gronberg BH, Benth JS, Baracos VE, Flotten O, Hjermstad MJ, Aass N, Jordhoy M. Low muscle mass is associated with chemotherapy-induced haematological toxicity in advanced non-small cell lung cancer. Lung Cancer. 2015 Oct;90(1):85-91. doi: 10.1016/j.lungcan.2015.07.001. Epub 2015 Jul 9. PMID 26198373
- [Background] de Jong C, Chargi N, Herder GJM, van Haarlem SWA, van der Meer F, van Lindert ASR, Ten Heuvel A, Brouwer J, de Jong PA, Devriese LA, Huitema ADR, Egberts TCG, de Bree R, Deneer VHM. The association between skeletal muscle measures and chemotherapy-induced toxicity in non-small cell lung cancer patients. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1554-1564. doi: 10.1002/jcsm.12967. Epub 2022 Mar 18. PMID 35301821
- See also: Danish Research Center for Equality in Cancer (COMPAS) homepage — https://www.sjaellandsuniversitetshospital.dk/afdelinger/onkologisk-afdeling-og-palliative-enheder/forskning/forskningsomraader/dansk-forskningscenter-for-lighed-i-kraeft-compas

DOCUMENTS (1):
  • Study Protocol (2026-02-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT06730685/Prot_000.pdf